CLINICAL TRIAL: NCT05822102
Title: Simultaneous quanTification of Elexacaftor/tezAcaftor/Ivacaftor Via Reverse Phase High Performance liquiD chromatographY
Acronym: STEADY
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS-3978
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis
Keywords: trikafta; elexacaftor/tezacaftor/ivacaftor (ETI); ETI; cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with Cystic Fibrosis who are taking ETI that has reached a steady state dosing level.: Blood samples will be collected from people with CF who are taking ETI at a continuous dosing regimen for a minimum of 14 days.

SUMMARY:
The purpose of this study is to support the clinical validation of a new assay to measure the levels of ivacaftor, tezacaftor, and elexacaftor (the components of Trikafta) in the bloodstream in order to achieve greater understanding of the effectiveness of this medication in all people with cystic fibrosis. Blood will be drawn at 3.0, 4.5, and 6.0 hours after taking the medication in the morning.

DETAILED DESCRIPTION:
Blood samples will be collected to measure steady state blood levels for participants who are being treated with elexacaftor/tezacaftor/ivacaftor (ETI). This study is being conducted to evaluate drug dosing in people with cystic fibrosis. The aim of this study is to support clinical validation of pharmacokinetics launch of the elexacaftor/tezacaftor/ivacaftor blood serum level assay to demonstrate instrument capabilities to pass ADx validation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from subject
* Diagnosis of CF
* Aged 18 years and older
* Use of ETI that has reached steady state dosing levels of ETI, defined as a continuous dosing regimen for a minimum of 14 days.

Exclusion Criteria:

* A person with CF (pwCF) that is either not taking ETI or dose not follow a continuous dosing regimen for a minimum of 14 days.
* Use of prohibited medications as outlined by package insert
* Pregnant or lactating people with CF
* Acute, severe deterioration in health requiring intensive care unit admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 100 people with CF who attend the Adult CF Program of Colorado at National Jewish Health and are actively taking ETI hat has reached steady state dosing levels of ETI (defined as a continuous dosing regimen for a minimum of 14 days) will be recruited and enrolled.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients with ETI in expected reference range | 3 hours, 4.5 hours and 6 hours after taking the medication
  Patient expected reference range determined by initial U.S FDA (2019 approval documentation): Cmax for Elexacaftor, Tezacaftor, Ivacaftor are 8.7± 2.1, 6.8 ± 1.5, 1.2 ± 0.3 mcg/mL, respectively. Limit of quantification estimated to be within +/- 20% of lowest calibration point of 0.2 mcg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Nick, MD, Principal Investigator — National Jewish Health
Locations (2):
- United States (2):
  - National Jewish Health, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No